CLINICAL TRIAL: NCT01251302
Title: Investigation of a Molecular Personalized Coronary Gene Expression Test on Cardiology Practice Pattern
Brief Title: Utility of a Molecular Personalized Coronary Gene Expression Test (Corus CAD or ASGES) on Cardiology Practice Pattern
Acronym: IMPACT-CARD
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000011; IMPACT-CARD (Other: CardioDx)
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Angina Pectoris; Coronary Artery Disease; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; CAD; CVD; CHD
Keywords: Corus CAD; Age/Sex/Gene Expression Score; Molecular Genetics; Atherosclerosis; ASGES; Gene Expression; GES; CAD; CVD; CHD; Clinical Utility; Precision Medicine; Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; IMPACT; IMPACT-CARD
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease; Chest Pain; Cardiovascular Diseases; Coronary Disease; Atherosclerosis; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — PaxGene tube for RNA collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective Cohort: Patient presenting with chest pain or anginal equivalent and receiving a resulted age, sex and gene expression score (ASGES) to assist in diagnosis.
  Interventions: Diagnostic Test: Corus CAD (ASGES)
- Retrospective Cohort: Patients presenting with chest pain or anginal equivalent who did not receive an age, sex and gene expression score (ASGES) to assist in diagnosis. Note: this cohort was historical.

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES) — Age/Sex/Gene Expression Score - ASGES
  Groups: Prospective Cohort

SUMMARY:
To investigate whether the use of Corus CAD (Age/Sex/Gene Expression score - ASGES) blood assay changes the diagnostic testing pattern in patients referred to a cardiologist for the evaluation of chest pain or anginal equivalent symptoms.

DETAILED DESCRIPTION:
A prospective cohort of 88 subjects receiving the Corus CAD (Age/Sex/Gene Expression score - ASGES) assay were compared to a retrospective cohort of 83 subjects that did not receive the assay.

ELIGIBILITY:
Inclusion Criteria:

1. Stable chest pain, typical or atypical angina or anginal equivalent
2. The patient has signed the appropriate Institutional Review Board approved Informed Consent Form.

Exclusion Criteria:

1. History of myocardial infarction
2. Current myocardial infarct (MI) or acute coronary syndrome
3. Current New York Heart Association (NYHA) class III or IV congestive heart failure symptoms
4. Any previous coronary revascularization
5. Any individuals with:

   1. Diabetes
   2. Suspected unstable angina
   3. Systemic infections
   4. Systemic inflammatory conditions
6. Any individuals currently taking:

   1. Steroids
   2. Immunosuppressive agents
   3. Chemotherapeutic agents
7. Recipient of any organ transplant

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll a patient population that present with chest pain or anginal equivalent symptoms who are referred to a cardiologist for evaluation.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in management practice pattern between preliminary and after Corus CAD (ASGES) decision | Up to 7 days
  Change in management pattern comparing the preliminary and after Corus CAD (ASGES) decision will be measured by the number of subjects with medical management downgrade or upgrade within the following predefined categories:
  1. No further cardiac testing or treatment
  2. Medical therapy for angina or non-cardiac chest pain
  3. Stress testing with or without imaging
  4. CT angiography
  5. Invasive cardiac catheterization
Change in management practice pattern between after Corus CAD decision and historical cohort. | up to 195 days
  Change in management pattern comparing the Corus CAD (ASGES) driven decision and the historical cohort ill be measured by the number of subjects with medical management downgrade or upgrade within the following predefined categories:
  1. No further cardiac testing or treatment
  2. Medical therapy for angina or non-cardiac chest pain
  3. Stress testing with or without imaging
  4. CT angiography
  5. Invasive cardiac catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, Study Director — CardioDx, Inc.
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] McPherson JA, Davis K, Yau M, Beineke P, Rosenberg S, Monane M, Fredi JL. The clinical utility of gene expression testing on the diagnostic evaluation of patients presenting to the cardiologist with symptoms of suspected obstructive coronary artery disease: results from the IMPACT (Investigation of a Molecular Personalized Coronary Gene Expression Test on Cardiology Practice Pattern) trial. Crit Pathw Cardiol. 2013 Jun;12(2):37-42. doi: 10.1097/HPC.0b013e3182822bd0. PMID 23680805